CLINICAL TRIAL: NCT04081844
Title: An Open-label, Multiple Dose, Fixed-sequence, 3-period Study to Evaluate the Pharmacokinetic and Pharmacodynamic Interactions Between HGP0904, HGP0608 and HCP1306 in Healthy Male Subjects
Brief Title: A Study to Evaluate the Pharmacokinetic and Pharmacodynamic Interactions Between HGP0904, HGP0608, and HCP1306 in Healthy Male Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HM-AMOS-101
Record Dates: First submitted 2019-09-02; First posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fixed-Sequence (Experimental): Period 1: Fasted state+HCP1306, Period 2: Fasted state+HGP0904+HGP0608, Period 3: Fasted state+HCP1306+HGP0904+HGP0608
  Interventions: Drug: HCP1306; Drug: HGP0904; Drug: HGP0608

INTERVENTIONS:
Drug: HCP1306 — Ezetimibe 10mg / Rosuvastatin 20mg (Rosuzet)
Drug: HGP0904 — Amlodipine 5mg(Norvasc)
Drug: HGP0608 — Losartan 100mg(Cozaar)

SUMMARY:
An Open-label, Multiple-dose, Fixed-sequence, 3-Period Study to Evaluate the Pharmacokinetic and Pharmacodynamic Interactions between HGP0904, HGP0608 and HCP1306 in Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Age 19~45 years in healthy volunteers
2. BMI is more than 18.5 kg/m^2 , no more than 29.9 kg/m^2
3. Subjects who agree to use medically accepted dual contraceptives up to two months after the last administration date of the clinical trial drug and not to provide sperm.
4. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
2. Subjects who judged ineligible by the investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Cmax,ss of Amlodipine | D18: pre-dose(0 hour), D26: pre-dose(0 hour), D27: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
AUCtau of Amlodipine | D18: pre-dose(0 hour), D26: pre-dose(0 hour), D27: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
Cmax,ss of Losartan | D18: pre-dose(0 hour), D26: pre-dose(0 hour), D27: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
AUCtau of Losartan | D18: pre-dose(0 hour), D26: pre-dose(0 hour), D27: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
Cmax,ss of EXP3174 | D18: pre-dose(0 hour), D26: pre-dose(0 hour), D27: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
AUCtau of EXP3174 | D18: pre-dose(0 hour), D26: pre-dose(0 hour), D27: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
Cmax,ss of Rosuvastatin | D1: pre-dose(0 hour), D5: pre-dose(0 hour), D6: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
AUCtau of Rosuvastatin | D1: pre-dose(0 hour), D5: dose(0 hour), D6: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
Cmax,ss of Free Ezetimibe | D1: pre-dose(0 hour), D5: dose(0 hour), D6: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
AUCtau of Free Ezetimibe | D1: pre-dose(0 hour), D5: dose(0 hour), D6: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
Cmax,ss of Total Ezetimibe | D1: pre-dose(0 hour), D5: dose(0 hour), D6: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
AUCtau of Total Ezetimibe | D1: pre-dose(0 hour), D5: dose(0 hour), D6: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation

SECONDARY OUTCOMES:
Cmin,ss of Amlodipine | D18: pre-dose(0 hour), D26: pre-dose(0 hour), D27: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
T max,ss of Amlodipine | D18: pre-dose(0 hour), D26: pre-dose(0 hour), D27: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
T1/2 of Amlodipine | D18: pre-dose(0 hour), D26: pre-dose(0 hour), D27: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
Cmin,ss of Losartan | D18: pre-dose(0 hour), D26: pre-dose(0 hour), D27: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
T max,ss of Losartan | D18: pre-dose(0 hour), D26: pre-dose(0 hour), D27: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
T1/2 of Losartan | D18: pre-dose(0 hour), D26: pre-dose(0 hour), D27: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
Cmin,ss of EXP3174 | D18: pre-dose(0 hour), D26: pre-dose(0 hour), D27: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
T max,ss of EXP3174 | D18: pre-dose(0 hour), D26: pre-dose(0 hour), D27: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
T1/2 of EXP3174 | D18: pre-dose(0 hour), D26: pre-dose(0 hour), D27: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
Cmin,ss of Rosuvastatin | D1: pre-dose(0 hour), D5: pre-dose(0 hour), D6: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
T max,ss of Rosuvastatin | D1: pre-dose(0 hour), D5: pre-dose(0 hour), D6: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
T1/2 of Rosuvastatin | D1: pre-dose(0 hour), D5: pre-dose(0 hour), D6: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
Cmin,ss of Free Ezetimibe | D1: pre-dose(0 hour), D5: dose(0 hour), D6: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
Tmax,ss of Free Ezetimibe | D1: pre-dose(0 hour), D5: dose(0 hour), D6: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
T1/2 of Free Ezetimibe | D1: pre-dose(0 hour), D5: dose(0 hour), D6: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
Cmin,ss of Total Ezetimibe | D1: pre-dose(0 hour), D5: dose(0 hour), D6: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
Tmax,ss of Total Ezetimibe | D1: pre-dose(0 hour), D5: dose(0 hour), D6: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation
T1/2 of Total Ezetimibe | D1: pre-dose(0 hour), D5: dose(0 hour), D6: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hour, D29: pre-dose(0 hour), D33: pre-dose(0 hour), D34: pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hour
  Pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Hospital (Anam), Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No